CLINICAL TRIAL: NCT00135850
Title: The Effect of Mobilized Stem Cell by G-CSF and VEGF Gene Therapy in Patients With Stable Severe Angina Pectoris
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gene G-CSF
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2002-10

CONDITIONS: Ischemic Heart Disease
Keywords: Gene therapy; VEGF; Stem cells; myocardial ischemia; angiogenesis
MeSH Terms: conditions — Myocardial Ischemia

INTERVENTIONS:
Genetic: VEGF-A165 plasmid

SUMMARY:
The aim of this study was to evaluate the mobilization of non-haematopoietic mesenchymal and haematopoietic stem cells from the bone marrow with granulocyte colony stimulating factor (G-CSF) treatment alone and in combination with vascular endothelial growth factor (VEGF) gene therapy in patients with severe chronic occlusive coronary artery disease.

DETAILED DESCRIPTION:
In recent clinical trials, vascular endothelial growth factor (VEGF) delivered as plasmid DNA percutaneously by a catheter-based, intramyocardial approach, have been demonstrated to be safe and to be associated with a reduction in angina and an increase in exercise time or an improvement in regional wall motion in "no-option patients" with chronic myocardial ischemia.

It has been demonstrated, that BM-derived stem cells mobilized by cytokines as granulocyte colony stimulating factor (G-CSF) were capable of regenerating the myocardial tissue, leading to improve the survival and cardiac function after myocardial infarction.

These data suggested that a combination therapy with exogenous administration of gene vascular growth factor combined with G-CSF mobilization of bone marrow stem cells might induce both angiogenesis and vasculogenesis in ischemic myocardium

ELIGIBILITY:
Inclusion Criteria:

* Reversible ischemia at an adenosine stress single photon emission computerized tomography (SPECT)
* A coronary arteriography demonstrating at least one main coronary vessel from which new collaterals/vessels could be supplied
* Age above 18 years
* Canadian Cardiovascular Society angina classification (CCS) > 3.

Exclusion Criteria:

* Ejection fraction <0.40
* Unstable angina pectoris
* Acute myocardial infarction within the last three months
* Diabetes mellitus with proliferative retinopathy
* Diagnosed or suspected cancer disease
* Chronic inflammatory disease
* Premenopausal women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2003-03; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Improvement in myocardial perfusion measured by single photon emission computerized tomography (SPECT)

SECONDARY OUTCOMES:
Clinical improvement

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, MD DMSc, Principal Investigator — Cardiac Catheterization Laboratory 2014, The Heart Centre, University Hospital, Rigshospitalet, DK-2100 Copenhagen Ø, Denmark
Locations (1):
- Cardiac Catheterization Laboratory 2014, The Heart Centre, University Hospital, Rigshospitalet, Copenhagen Ø, Denmark